CLINICAL TRIAL: NCT02656498
Title: An Open Label, Multicenter Study for Evaluation of the Clinical Utility of [18F]THK-5351 Positron Emission Computed Tomography in Cognitively Healthy Volunteers, Subjects With Mild Cognitive Impairment, Subjects With Alzheimer's Disease and Subjects With Other Neurodegenerative Diseases
Brief Title: [18F]THK-5351 Positron Emission Computed Tomography Study of Normal, Mild Cognitive Impairment, Alzheimer's Disease and Other Neurodegenerative Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jae Seung Kim (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jae Seung Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: THK-15002
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Neurodegenerative Diseases
Keywords: Tau, neurodegeneration, positron emission computed tomography
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurodegenerative Diseases; Pick Disease of the Brain; Nerve Degeneration | interventions — THK5351

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitively Healthy Subjects (Experimental): Cognitively healthy subjects will receive an IV injection, [18F]THK-5351 at baseline and also receive an IV injection, [18F]THK-5351 at 24 months.
  Interventions: Drug: [18F]THK-5351
- MCI Subjects (Experimental): MCI Subjects will receive an IV injection, [18F]THK-5351 at baseline and also receive an IV injection, [18F]THK-5351 at 24 months.
  Interventions: Drug: [18F]THK-5351
- AD Subjects (Experimental): AD Subjects will receive an IV injection, [18F]THK-5351 at baseline and also receive an IV injection, [18F]THK-5351 at 24 months.
  Interventions: Drug: [18F]THK-5351
- Subjects with other neurodegenerative disease (Experimental): Subjects with other neurodegenerative disease will receive an IV injection, [18F]THK-5351 at baseline.
  Interventions: Drug: [18F]THK-5351

INTERVENTIONS:
Drug: [18F]THK-5351 — Imaging for evaluating the accumulation of abnormal tau protein in the brain
  Other Names: FluoroTau

SUMMARY:
This is a cross-sectional and longitudinal study to evaluate the clinical utility of [18F]THK-5351 positron emission computed tomography in cognitively healthy volunteers, mild cognitive impairment (MCI), Alzheimer's disease (AD) and other neurodegenerative patients.

ELIGIBILITY:
Inclusion Criteria:

1. General Subject Inclusion Criteria

   In order to be eligible for participation in this trial, the subject must:
   * Be ≥ 40 and < 80 years of age at the Screening Visit.
   * Be able to read at a 6th grade level or equivalent, (as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.)
   * Be able to speak, read, hear, and understand the language of the trial staff, and the informed consent form, and possess the ability to respond verbally to questions, follow instructions, and complete questionnaires and detailed neuropsychological test.
   * Have results of clinical laboratory tests/physical examination, vital signs, and ECG within normal limits (at 90 days prior to [18F]THK-5351 positron emission computed tomography) or clinically acceptable to the investigator at screening.
   * Be able to possess the ability to respond verbally to questions, follow instructions, and underwent research assessment, including brain images based on the investigator's judgment. Each subject is also able and willing to adhere visit schedules.
   * If female, not be of childbearing potential as indicated by one of the following
   * Each subject (or legal representative) must sign the informed consent form in accordance with local requirements after the scope and nature of the investigation have been explained to them, and before screening assessments.
   * Each subject must be willing to provided blood samples for genotyping apolipoprotein E
2. Cognitively Healthy Subjects
3. MCI Subjects
4. AD Subjects
5. Subjects with other neurodegenerative disease

Exclusion Criteria

The subject must be excluded from participating in the trial if the subject fulfil any single criteria described below:

1. General Exclusion Criteria

* Based on the investigators' judgement, if the patient is not capable of communicating with the site personnel, if the patient is not proficient in the language in which the psychometric tests will be completed, or if the patient is not sufficient for compliance with the study procedures.
* The patient has an abnormal physical examination or abnormal laboratory test results at the screening that are clinically significant to affect results of the research, as judged by the investigator.
* If the patient has or is suspicious of having a hypersensitivity or allergy to [18F] THK-5351 or its derivatives.
* The patient is pregnant, is attempting to become pregnant, or is nursing (breast-feeding) children.
* The patient has a history of alcoholism or drug dependency/abuse within the last 2 years before screening.
* The patient has contraindications to undergo positron emission computed tomography or MRI, which include but are not restricted to the examples below: claustrophobia, cardiac pacemaker, metal devices around the eye or spinal cord, cochlear implant, etc.) at the screening visit.
* The patient has been treated with any investigational medicinal product (IMP) within 30 days prior to the screening visit.
* The patient has been tested positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), HIV Antibody, or syphilis serum test at the screening visit.
* The patient has been receiving an anti-cholinergic drug in a regular basis within 3 months prior to the screening visit.
* The patient has evidence of a clinically relevant neurological disorders other than the disease being studied (i.e., prodromal AD) at screening, including but not limited to: territorial cerebral infarction, intracranial hemorrhage, multiple sclerosis, neurosyphilis, mental retardation, hypoxic encephalopathy, major head trauma with loss of consciousness that led to persistent cognitive deficits.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Cross-sectional [18F]THK-5351 Imaging Results | 50-70 minutes post injection
  Compare Standard uptake value ratio (SUVR) and distribution of [18F]THK-5351 in subjects with MCI, subjects with AD, subjects with other neurodegenerative disease and cognitively healthy individuals.
Assess the rate of change of tau deposition as measured by [18F]THK-5351 uptake (SUVR) over time | 24 months
  Compare Standard uptake value ratio (SUVR) and distribution of [18F]THK-5351 in subjects with MCI, subjects with AD, subjects with other neurodegenerative disease and cognitively healthy individuals.

SECONDARY OUTCOMES:
Correlation between standard uptake value ratio (SUVR) of [18F]THK-5351 positron emission computed tomography and neuropsychiatric test scores | 50-70 minutes post-injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]THK-5351 positron emission computed tomography and scores of neuropsychiatric test
Correlation between standard uptake value ratio (SUVR) of [18F]THK-5351 positron emission computed tomography and indices of structural MRI | 50-70 minutes post-injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]THK-5351 positron emission computed tomography and indices of structural MRI including cortical thickness, hippocampal atrophy.
Correlation between standard uptake value ratio (SUVR) of [18F]THK-5351 positron emission computed tomography and indices of functional MRI | 50-70 minutes post-injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]THK-5351 positron emission computed tomography and indices of functional MRI derived from diffusion tensor imaging and resting state functional MRI.
Correlation between standard uptake value ratios (SUVR) and distribution of [18F]THK-5351 positron emission computed tomography and amyloid positron emission computed tomography | 50-70 minutes post-injection
  We will evaluate correlation between standard uptake value ratio (SUVR) and distribution of [18F]THK-5351 positron emission computed tomography and those of amyloid positron emission computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Kim, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Chun MY, Lee J, Jeong JH, Roh JH, Oh SJ, Oh M, Oh JS, Kim JS, Moon SH, Woo SY, Kim YJ, Choe YS, Kim HJ, Na DL, Jang H, Seo SW. 18F-THK5351 PET Positivity and Longitudinal Changes in Cognitive Function in beta-Amyloid-Negative Amnestic Mild Cognitive Impairment. Yonsei Med J. 2022 Mar;63(3):259-264. doi: 10.3349/ymj.2022.63.3.259. PMID 35184428
- [Derived] Park JE, Yun J, Kim SJ, Shim WH, Oh JS, Oh M, Roh JH, Seo SW, Oh SJ, Kim JS. Intra-individual correlations between quantitative THK-5351 PET and MRI-derived cortical volume in Alzheimer's disease differ according to disease severity and amyloid positivity. PLoS One. 2019 Dec 13;14(12):e0226265. doi: 10.1371/journal.pone.0226265. eCollection 2019. PMID 31834916